CLINICAL TRIAL: NCT03160846
Title: Inotrope, Evaluation and Research (INTERPRET) Patient Registry Program
Brief Title: The Inotrope Evaluation and Research Patient Registry
Acronym: INTERPRET
Status: Completed | Type: Observational
Sponsor: Coram Clinical Trials (Other)
Collaborators: Columbia University (Other); Northwestern University (Other); University of Kansas Medical Center (Other); University of Alabama at Birmingham (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: CT-10-05
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
Keywords: Inotrope; Milrinone; Dopamine; Dobutamine
MeSH Terms: conditions — Heart Failure | interventions — Milrinone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Inotrope — Home intravenous infusion of Dobutamine, Dopamine, or Milrinone
  Other Names: Primacor

SUMMARY:
The INTERPRET Inotrope Evaluation and Research Patient Registry is a longitudinal, observational study designed to look at the demographics and outcomes of heart failure patients on inotropic therapy administered in the home or infusion suite setting. The data gathered in this registry will provide information on how a patient's quality of life and symptoms change over time while on inotrope therapy, and help healthcare providers to have a better understanding of the benefits and risks associated with bridge-to-treatment and palliative care.

DETAILED DESCRIPTION:
Eligible patients will be consented by the site investigator or staff to participate in the Registry at the time of referral for home care. Clinical data, including dosing, symptom severity, lab values, and hospitalizations, along with data on quality-of-life and patient compliance with treatment, will be collected by the home care nurses and pharmacists. The Registry's goal is to significantly contribute to the medical understandings of heart failure treatment and to improve the quality of care for heart failure patients in the United States through active publication of registry findings and disease management approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be prescribed inotropic treatment (milrinone, dobutamine or dopamine)
* Patient must be referred to Coram for this treatment in an alternate site of care, either home or infusion suite
* Patient must be willing to receive care and comply with the teaching and training necessary to administer treatment
* Patient is age 18 or over

Exclusion Criteria:

* Patient is unable to start, or stops taking, inotropic medication
* Patient and/or patient insurance will not cover cost of home inotropic treatment with Coram, or patient elects not to start treatment
* Patient is under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified by investigator and study staff from among patients admitted to hospital for HF that are being discharged to receive inotropic therapy in the home or infusion suite.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Mean time of survival post-treatment | Through study completion, on average 6 months
  Recording length of time on treatment (in days) from start of care at Coram to study discharge date
Number of re-hospitalizations | Through study completion, on average 6 months
  Recorded on the Pharmacy Clinical Progress Report
Duration of re-hospitalizations | Through study completion, on average 6 months
  The duration (days) of re-hospitalization visits
Primary cause of re-hospitalization visits | Through study completion, on average 6 months
  The primary cause of re-hospitalization visits following treatment will be recorded by nurse on patient clinical progress report from a drop-down list with the following options: Central venous access device malfunction, central venous access device infection, cognitive changes, fatigue, dyspnea, fever, chest pain, blood pressure instability, edema, weight gain, nausea and anorexia, and other
Implantable cardioverter defibrillator (ICD) activity | Weekly, through study completion (an average of 6 months)
  Number of ICD firings as recorded by nurse on patient clinical progress report
Patient reported symptom severity questionnaire | Monthly, through study completion (an average of 6 months)
  A patient completed questionnaire will be used to report the severity of the following symptoms: Pain, Fatigue, Edema, Shortness of breath (with exertion), Shortness of breath (without exertion)
Quality of life assessment: Questionnaire | Monthly, through study completion (an average of 6 months)
  The patient completed Kansas City Cardiomyopathy Questionnaire will be used to report the overall patient quality of life

SECONDARY OUTCOMES:
Concomitant medication use | Weekly, through study completion (an average of 6 months)
  Patient medication profiles will be monitored for presence or absence of additional medications other than inotropes
Additional patient symptoms | Weekly, through study completion (an average of 6 months)
  A weekly nurse completed clinical progress report will record the presence or absence of the following: increased urination at night, swollen abdomen, breathing problem when lying down to sleep, cough with frothy sputum, loss of appetite, depression, and confusion and/or memory challenges

CONTACTS AND LOCATIONS:
Overall Officials: Erica Blanchard, PharmD, Study Director — Coram/CVS specialty infusion
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, Bluhm Cardiovascular Institute, Chicago, Illinois
  - The University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center/Vivian and Seymour Milstein Family Heart Center, New York, New York

REFERENCES:
- [Result] Checkley et. al. CONTINUOUS HOME INTRAVENOUS INOTROPIC THERAPY DECREASES SYMPTOM SEVERITY AND MAY REDUCE HOSPITALIZATIONS IN PATIENTS WITH ADVANCED HEART FAILURE Journal of the American College of Cardiology Mar 2018, 71 (11 Supplement) A806; DOI: 10.1016/S0735-1097(18)31347-0